CLINICAL TRIAL: NCT01606540
Title: The Influence of Non-steroid Antiinflammatory Drugs (NSAID) to Heal Colles Fracture.
Brief Title: Non-steroid Antiinflammatory Drugs to Heal Colles Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: N-20120015
Record Dates: First submitted 2012-05-15; First posted 2012-05-25 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Colles Fracture
Keywords: Colles fracture; Non-steroid antiinflammatory drugs; Bone healing
MeSH Terms: conditions — Colles' Fracture | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reposition and immobilism (Experimental): The patient are under sedation before reposition. The patient will be injected with 8-10 ml 1% Lidocain.
  After reposition the patient is asked to fill in a questionnaire with information of experienced pain based on VAS score. The patient note down the experience of pain each day 14 days after reposition.
  Interventions: Drug: Tablets Ibumetin and placebo
- Surgery (Active Comparator): The method of surgery is type bridging.
  After surgery the patient is asked to fill in a questionnaire with information of experienced pain based on VAS score. The patient note down the experience of pain each day 14 days after operation.
  Interventions: Drug: Tablets Ibumetin and placebo

INTERVENTIONS:
Drug: Tablets Ibumetin and placebo — Group A: Daily tablets Ibumetin, 600 mg x 3, 7 days after reposition.
  Group B: Daily tablets Ibumetin, 600 mg x 3, 3 days after reposition. The following days placebo tablets.
  Group C: Placebo tablets 1 week after reposition.
  Other Names: No other names.
  Arms: Reposition and immobilism
Drug: Tablets Ibumetin and placebo — Group A: Daily tablets Ibumetin, 600 mg x 3, 7 days after surgery.
  Group B: Daily tablets Ibumetin, 600 mg x 3, 3 days after surgery. The following days placebo tablets.
  Group C: Placebo tablets for 1 week after surgery.
  Other Names: No other names.
  Arms: Surgery

SUMMARY:
It is believed that some painkillers (NSAID drugs) slow bone healing but the knowledge is based only on experimental studies with animals whose results are automatically translated for humans. The purpose is to examine whether these drugs slow bone healing and what relationship there is between different bone examinations, scan for osteoporosis, bone marker laboratory tests, radiological controls and histology of newly formed bone under a microscope.

DETAILED DESCRIPTION:
One of the most popular painkillers in the world is known as NSAID (non-steroidal anti-inflammatory drugs). Many studies with animals have been made which show a clear tendency for delayed bone healing by taking NSAIDs.

It is known that an early intake of NSAIDs prevents ectopic ossification in patients, receiving total hip prosthesis. However, cases of prosthetic loosening and instability after 10 years were almost exclusively observed in the group of patients who received NSAIDs postoperatively. However, very few clinical studies still show this tendency. In this study we include patients with fresh fracture in the wrist; Colles fracture. The fracture may seem unstable when there is a lack of bone healing. These fractures are very common in the orthopaedic clinic.

Although there is no dislocation of the fragments, newly formed bone can be weaker as demonstrated by DEXA scanning (bone mineral density measurement). Histological examination of the healing bone can give a definitive answer whether the bone was affected or not. Thus, the possibilities of studying NSAIDs affect on bone healing in humans and the clinical significance are very positive.

ELIGIBILITY:
Inclusion Criteria:

* Patients giving written informed consent and authority
* Patients with Colles fracture who require surgery by means of an external fixation or type bridging with or without suture.
* Patients who clinically and radiographically are diagnosed for reposition and therefore require external fixation or type bridging with or without suture.

Exclusion Criteria:

* Patients who have been given adrenal cortex hormone.
* Patients who have been given non-steroid antiinflammatory drugs (NSAID).
* Patients who have not been giving written informed consent and authority.
* Patients who smoke more than 20 cigarettes daily.
* Patients who consume more than 14 drinks weekly.
* Lack of mental and physical ability to follow the directions according to the protocol.
* Medical contraindication to non-steroid antiinflammatory drugs.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-06; Primary Completion 2020-03-20 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of dislocation. | An expected average of 5 weeks
  By means of new radiographic technology the investigator is able to determine the difference between any migration of fragments precisely.

SECONDARY OUTCOMES:
Pain score by VAS scale. | An expected average of 2 weeks.
  Every patient keeps a pain log 2 weeks after surgery.
Bone Mineral Density. | An expected average of 3 months
  By means of DEXA scanning the bone mineral density will be evaluated.
Movement deflections. | An expected average of 5 weeks
  Evaluation of flexion, extension, pronation and supination after 1 week, 2 weeks, 6 weeks and 3 months.
  DASH score after 3 months and 1 year.
Predictors for bone healing. | An expected average of 3 months
  To determine the predictors for bone healing in cooperation with Immunodiagnostic Systems.
Determine ossification. | An expected average of 3 months
  To perform a core biopsi in order to determinating ossification of callus.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Aliuskevicius, M.D., Principal Investigator — Orthopaedic Research Unit, Aalborg University Hospital
Locations (1):
- Orthopaedic Surgery Research Unit, Aalborg University Hospital, Aalborg, Denmark